CLINICAL TRIAL: NCT05359315
Title: An Open Prospective Observational Study Evaluating the Efficacy and Tolerability of Interferon Gamma (Ingaron) Injections in Patients With Drug-resistant Pulmonary Tuberculosis
Brief Title: Study on the Use of Interferon Gamma (Ingaron) Injections in Patients With Drug-resistant Pulmonary Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: STING-2021
Record Dates: First submitted 2022-04-22; First posted 2022-05-03 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Tuberculosis
Keywords: treatment of drug-resistant pulmonary tuberculosis; interferon gamma; drug resistant
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Interferon-gamma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Ingaron + basic TB therapy 500,000 IU once daily for 3 months followed by 3 months follow-up
  Interventions: Drug: Interferon-Gamma
- No Intervention: only basic anti-tuberculosis therapy

INTERVENTIONS:
Drug: Interferon-Gamma — received by microbiological synthesis; specific antiviral activity on cells is 2x10*7 Units per mg of protein
  Other Names: Ingaron; Interferon gamma human recombinant
  Groups: Experimental

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of the complex therapy of drug-resistant respiratory tuberculosis using the drug Ingaron, a lyophilisate for the preparation of a solution for injection for intramuscular or subcutaneous administration of 500,000 IU.

DETAILED DESCRIPTION:
Open prospective observational cohort study. During the recruitment phase, a preliminary assessment of eligibility and non-inclusion criteria will be carried out.

Subject to prior compliance with all inclusion criteria and none of the exclusion criteria, after signing a voluntary informed consent, the patient will be included in the study.

Patients will be divided into groups, depending on the therapy prescribed to them as part of routine clinical practice (according to clinical guidelines):

Group 1:

Pathogenetic therapy with the use of the drug Ingaron + basic anti-tuberculosis therapy in accordance with approved clinical guidelines.

Group 2:

Basic anti-tuberculosis therapy in accordance with approved clinical guidelines.

When a patient is included in the study (Visit 0), an initial examination will be carried out, in accordance with generally accepted principles of treatment monitoring, which includes: history taking, physical examination, registration of vital signs, ECG, blood samples for general clinical, biochemical analysis, general analysis urine, bacteriological examination by sputum smear microscopy and sputum culture on dense nutrient media with drug sensitivity assessment, computed tomography and chest radiography.

The inclusion/exclusion criteria will be checked. The expected duration of the study for each patient will be no more than 204 days.

After the start of therapy, patients will be recorded monthly with physical examination data with registration of vital signs, general clinical, biochemical analyzes, urinalysis, smear microscopy and sputum culture. X-ray examination and clinical evaluation of effectiveness will be carried out every 2 months. At visit 7 (after 6 months from the start of therapy), an evaluation of computed tomography and chest x-ray in dynamics with an assessment of the effectiveness of therapy, as well as ECG, physical examination with registration of vital signs, general clinical, biochemical analyzes, general urinalysis, smear microscopy and culture of sputum.

At visits 1, 4 and 7 immunological parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women 18-75 years of age.
* For women of childbearing age who are fertile: Agree to completely abstain from sexual intercourse or use dual methods of contraception to prevent pregnancy while participating in the study.
* Verified diagnosis of pulmonary tuberculosis (infiltrative tuberculosis, fibrous-cavernous tuberculosis in the infiltration phase).
* A positive sputum smear microscopy test result for acid-fast bacterium, assessed as moderate (++) or massive bacterial excretion (+++) no earlier than 30 days prior to enrollment in the study.
* Established resistance of the isolated pathogen to at least rifampicin, determined by molecular genetic or cultural methods for determining drug susceptibility.
* Prescribing the current baseline chemotherapy regimen according to clinical guidelines no earlier than 14 days prior to enrollment in the study.
* Compliance with prescribed therapy.
* No concomitant immunotherapy, or 6 months from the last dose of an immunomodulatory drug to the start of therapy.
* Absence of comorbidities and therapy that may affect the interpretation of study results, in the opinion of the investigator.
* Signed written informed consent to participate in the study.
* Willingness and ability to follow protocol requirements throughout the study.

Exclusion Criteria:

* For women: pregnant, breastfeeding or planning a pregnancy during the study period.
* Caseous pneumonia.
* Asthma, with the exception of mild intermittent asthma.
* Systemic fungal infections.
* Use of any investigational drug within 30 days prior to screening.
* Oncological diseases (cytotoxic chemotherapy, current or received within the last 3 months before the start of treatment).
* Chronic diseases of the liver or kidneys (an increase in liver transaminases more than 5 times the upper limit of laboratory norms for these indicators; an increase in creatinine above 2 mg / 100 ml (or μmol / l)).
* Diabetes.
* HIV infection or other immunodeficiency conditions.
* Inability, in the opinion of the investigator, to comply with the treatment regimen and the requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with drug-resistant pulmonary tuberculosis with bacterial excretion
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Sputum smear conversion according to microscopy. | 1 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 1 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion according to microscopy. | 2 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 2 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion according to microscopy. | 3 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 3 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion according to microscopy. | 4 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 4 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion according to microscopy. | 5 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 5 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion according to microscopy. | 6 months
  Sputum smear conversion according to microscopy. Percentage of patients.
Sputum smear conversion according to microscopy. | 6 months
  Sputum smear conversion according to microscopy. Mean time to clinical response.
Sputum smear conversion by culture. | 1 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 1 months
  Sputum smear conversion by culture. Mean time to clinical response.
Sputum smear conversion by culture. | 2 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 2 months
  Sputum smear conversion by culture. Mean time to clinical response.
Sputum smear conversion by culture. | 3 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 3 months
  Sputum smear conversion by culture. Mean time to clinical response.
Sputum smear conversion by culture. | 4 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 4 months
  Sputum smear conversion by culture. Mean time to clinical response.
Sputum smear conversion by culture. | 5 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 5 months
  Sputum smear conversion by culture. Mean time to clinical response.
Sputum smear conversion by culture. | 6 months
  Sputum smear conversion by culture. Percentage of patients.
Sputum smear conversion by culture. | 6 months
  Sputum smear conversion by culture. Mean time to clinical response.

SECONDARY OUTCOMES:
The effectiveness of therapy according to X-ray examination of the chest. | 2 months
  The effectiveness of therapy according to X-ray examination of the chest. Percentage of patients.
The effectiveness of therapy according to X-ray examination of the chest. | 4 months
  The effectiveness of therapy according to X-ray examination of the chest. Percentage of patients.
The effectiveness of therapy according to X-ray examination of the chest. | 6 months
  The effectiveness of therapy according to X-ray examination of the chest. Percentage of patients.
The effectiveness of therapy according to computed tomography of the chest. | 6 months
  The effectiveness of therapy according to computed tomography of the chest. Percentage of patients.
The effectiveness of therapy according to clinical examination. | 2 months
  The effectiveness of therapy according to clinical examination. Average score. The dynamics of clinical symptoms will be determined based on an assessment of the severity of intoxication (general) symptoms and respiratory complaints according to a 4-point system, where the minimum score is 0 - absent, the maximum 3 - pronounced
The effectiveness of therapy according to clinical examination. | 4 months
  The effectiveness of therapy according to clinical examination. Average score. The dynamics of clinical symptoms will be determined based on an assessment of the severity of intoxication (general) symptoms and respiratory complaints according to a 4-point system, where the minimum score is 0 - absent, the maximum 3 - pronounced
The effectiveness of therapy according to clinical examination. | 6 months
  The effectiveness of therapy according to clinical examination. Average score. The dynamics of clinical symptoms will be determined based on an assessment of the severity of intoxication (general) symptoms and respiratory complaints according to a 4-point system, where the minimum score is 0 - absent, the maximum 3 - pronounced
Change in immunological status (CD4 and CD8 lymphocyte populations) compared with baseline values (before therapy). | 3 months
  Change in immunological status (CD4 and CD8 lymphocyte populations) compared with baseline values (before therapy). Averages.
Change in immunological status (CD4 and CD8 lymphocyte populations) compared with baseline values (before therapy). | 6 months
  Change in immunological status (CD4 and CD8 lymphocyte populations) compared with baseline values (before therapy). Averages.
Mortality rate. | 6 months
  Mortality rate. The proportion of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- FSBI "NMIC FPI" of the Ministry of Health of Russia, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No